CLINICAL TRIAL: NCT01285752
Title: A Study of AK106-001616 in Patients With Rheumatoid Arthritis (RA)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Asahi Kasei Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AK106 II-02
Record Dates: First submitted 2011-01-27; First posted 2011-01-28 (Estimated); Last update posted 2016-07-25 (Estimated); Status verified 2012-04

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — AK106-001616

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- 1 (Experimental)
  Interventions: Drug: AK106-001616
- 2 (Experimental)
  Interventions: Drug: AK106-001616
- 3 (Active Comparator)
  Interventions: Drug: Active comparator

INTERVENTIONS:
Drug: AK106-001616
  Arms: 1
Drug: AK106-001616
  Arms: 2
Drug: Active comparator
  Arms: 3

SUMMARY:
To investigate the efficacy and safety of AK106-001616 in patients with rheumatoid arthritis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of RA (class I to III)
* Stable dose of methotrexate (at least 12 weeks)

Exclusion Criteria:

* Pregnant or breastfeeding
* Abnormal screening laboratory test values considered to be clinically significant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2011-02; Primary Completion 2012-01 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (26):
- Czechia (5):
  - Hlučín
  - Hostivice
  - Prague
  - Uherské Hradiště
  - Zlín
- Germany (3):
  - Berlin
  - Frankfurt
  - Hamburg
- Hungary (3):
  - Balatonfüred
  - Budapest
  - Debrecen
- Poland (5):
  - Bialystok
  - Elblag
  - Lublin
  - Poznan
  - Warsaw
- Slovakia (2):
  - Bratislava
  - Martin
- Ukraine (6):
  - Donetsk
  - Kharkiv
  - Kyiv
  - Ternopil
  - Vinnytsa
  - Zaporizhzhia
- United Kingdom (2):
  - Cambridge
  - Sheffield